CLINICAL TRIAL: NCT00680914
Title: Primary Vaccination Course in Children Receiving the Pneumococcal Vaccine GSK 1024850A or Prevenar™ Co-administered With Hiberix™
Brief Title: Primary Vaccination Course in Children Receiving Pneumococcal Conjugate Vaccine GSK 1024850A or Prevenar™ and Hiberix™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 110808
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2010-06-14 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Infections, Streptococcal
Keywords: Streptococcus pneumoniae; pneumococcal conjugate vaccine
MeSH Terms: conditions — Streptococcal Infections | interventions — PHiD-CV vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Synflorix Group (Experimental): Subjects received 3 doses of Synflorix vaccine co-administered with Hiberix vaccine at Study Months 0, 2 and 4.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A (Synflorix); Biological: GSK Biologicals' Hiberix™
- Prevenar Group (Active Comparator): Subjects received 3 doses of Prevenar vaccine co-administered with Hiberix vaccine at Study Months 0, 2 and 4.
  Interventions: Biological: Prevenar; Biological: GSK Biologicals' Hiberix™

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A (Synflorix) — 3 doses administered intramuscularly.
  Arms: Synflorix Group
Biological: Prevenar — 3 doses administered intramuscularly.
  Arms: Prevenar Group
Biological: GSK Biologicals' Hiberix™ — 3 doses administered intramuscularly.
  Other Names: Hib

SUMMARY:
The purposes of this study are:

To demonstrate the immunogenicity in terms of antibody response following primary vaccination of Korean infants with the pneumococcal conjugate vaccine GSK 1024850A compared to Prevenar™ when co-administered with a Haemophilus influenzae type b (Hib) vaccine in children during the first 6 months of life.

To evaluate the safety/reactogenicity in terms of solicited and unsolicited symptoms and serious adverse events following primary vaccination of Korean infants with the pneumococcal conjugate vaccine GSK 1024850A.

DETAILED DESCRIPTION:
Vaccination course at 2, 4, 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including 6-12 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol should be enrolled in the study.
* Written and signed informed consent obtained from the parent(s)/guardian(s) of the child/ward.
* Free of any known or suspected health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive, with a birth weight of at least 2.5 kilogram.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of the study vaccines, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not allowed by the study protocol during the study period. Vaccines included in the Korean routine immunization schedule can be administered at least one week before or at least one month after the administration of the study vaccines. Recommended live vaccines not included in the Korean routine immunization schedule can be given at least one month before or at least one month after the administration of the study vaccines.
* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period (Hepatitis B immunoglobulins at birth are allowed).
* Previous vaccination against Streptococcus pneumoniae and/or Haemophilus influenzae type b.
* History of, or intercurrent Streptococcus pneumoniae and/or Haemophilus influenzae type b disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment. Study entry should be delayed until the illness has improved.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 503 (Actual)
Dates: Start 2008-06-10 (Actual); Primary Completion 2009-05-08 (Actual); Study Completion 2009-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- South Korea (11):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gyeongnam
  - GSK Investigational Site, Iksan
  - GSK Investigational Site, Jeju City
  - GSK Investigational Site, Jeonju Jeonbuk
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
  - GSK Investigational Site, Wonju-si Kangwon-do

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kim CH, Kim JS, Cha SH, Kim KN, Kim JD, Lee KY, Kim HM, Kim JH, Hyuk S, Hong JY, Park SE, Kim YK, Kim NH, Fanic A, Borys D, Ruiz-Guinazu J, Moreira M, Schuerman L, Kim KH. Response to primary and booster vaccination with 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine in Korean infants. Pediatr Infect Dis J. 2011 Dec;30(12):e235-43. doi: 10.1097/INF.0b013e31822a8541. PMID 21817957
- [Background] Kim CH et al. Immunogenicity and safety of 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Korean children. Abstract presented at the Korean Society of Pediatric Infectious Diseases - 2011 Spring Conference. Seoul, South Korea, 7-11 June 2011.
- [Background] Kim CH et al. Immunogenicity of a 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHiD-CV) and co-administered vaccines following primary vaccination in Asian infants. Abstract presented at the 5th Asian Congress of Pediatric Infectious Diseases (ACPID). Taipei, Taiwan, 23-26 September 2010.
- [Background] Kim JS et al. Safety and reactogenicity of primary vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Korean infants. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Kim KH et al. Immunogenicity of primary vaccination with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Korean infants. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L, Wysocki J, Tejedor JC, Knuf M, Kim KH, Poolman J. Prediction of pneumococcal conjugate vaccine effectiveness against invasive pneumococcal disease using opsonophagocytic activity and antibody concentrations determined by enzyme-linked immunosorbent assay with 22F adsorption. Clin Vaccine Immunol. 2011 Dec;18(12):2161-7. doi: 10.1128/CVI.05313-11. Epub 2011 Oct 12. PMID 21994351
- [Background] Schuerman L et al. Immune responses against cross-reactive pneumococcal serotypes 6A and 19A with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. OPA assay is more reliable predictor of vaccine effectiveness against invasive pneumococcal disease (IPD) than ELISA antibody measurements. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Population variability in antibody responses following pneumococcal conjugate vaccination: experience with the non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Population variability of opsonophagocytic activity following 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate (PHiD-CV) vaccination more limited than antibody responses. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110808 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synflorix Group | Prevenar Group
Started | 374 | 129
Completed | 364 | 125
Not Completed | 10 | 4
Not completed — Consent withdrawal | 6 | 3
Not completed — Lost to Follow-up | 4 | 0
Not completed — serious adverse event (SAE) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix Group | Prevenar Group | Total
Number analyzed (Participants) | 374 | 129 | 503
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (1.49) | 9.5 (1.43) | 9.5 (1.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 71 | 260
  Male | 185 | 58 | 243
Region of Enrollment [Number; unit: participants]
  East Asia | 373 | 129 | 502 (0) [0 to 0]
  Southeast Asia | 1 | 0 | 1 (0) [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Pneumococcal Serotypes Antibody Concentrations Above the Cut-Off Value
Description: Anti-pneumococcal antibody cut-off value assessed was 0.20 microgram per milliliter (ug/mL).
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after administration of 3rd dose of the pneumococcal conjugate vaccine
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 344 | 123
subjects
  Anti-1 | 344 | 7
  Anti-4 | 343 | 123
  Anti-5 | 344 | 18
  Anti-6B | 318 | 121
  Anti-7F | 344 | 4
  Anti-9V | 343 | 122
  Anti-14 | 342 | 123
  Anti-18C | 343 | 123
  Anti-19F | 340 | 123
  Anti-23F | 331 | 121

2. Secondary Outcome: Number of Subjects With a Seropositivity Status Against Protein D and Defined Pneumococcal Serotypes
Description: Seropositivity status for protein D is defined as anti protein D (anti-PD) antibody concentrations >= 100 Enzyme-Linked Immuno Sorbent Assay (EL) units EL.U/mL.
  Seropositivity status for pneumococcal serotypes is defined as anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations >= 0.05 ug/mL.
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 344 | 123
subjects
  Anti-PD | 343 | 123
  Anti-1 | 344 | 44
  Anti-4 | 344 | 123
  Anti-5 | 344 | 85
  Anti-6B | 337 | 122
  Anti-7F | 344 | 22
  Anti-9V | 343 | 123
  Anti-14 | 344 | 123
  Anti-18C | 344 | 123
  Anti-19F | 344 | 123
  Anti-23F | 340 | 122

3. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Pneumococcal Serotypes Contained in the Vaccine Above the Cut-off Value
Description: The results were presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. In this assay the cut-off value for opsonophagocytic activity against pneumococcal antibody assessed was >= 8.
  The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available data.
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 165 | 63
subjects
  Opsono-1 (N=162; 62) | 150 | 8
  Opsono-4 (N=161; 63) | 158 | 63
  Opsono-5 (N=165; 62) | 161 | 6
  Opsono-6B (N=162; 63) | 152 | 63
  Opsono-7F (N=164; 59) | 164 | 40
  Opsono-9V (N= 165; 63) | 164 | 62
  Opsono-14 (N= 165; 63) | 163 | 62
  Opsono-18C (N= 159; 63) | 142 | 61
  Opsono-19F (N=164; 61) | 159 | 55
  Opsono-23F (N= 164; 63) | 160 | 62

4. Secondary Outcome: Number of Subjects With Cross-reactive Pneumococcal Serotype Antibody Concentrations Above the Cut-Off Value
Description: Anti-pneumococcal antibody cut-off value assessed was 0.20 microgram per milliliter (ug/mL).
  Pneumococcal cross-reactive serotypes were 6A and 19A.
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 344 | 123
subjects
  Anti-6A | 232 | 85
  Anti-19A | 203 | 33

5. Secondary Outcome: Antibody Concentrations Against Pneumococal Serotypes Contained in the Vaccine
Description: Concentrations are reported as Geometric Mean Concentrations in ug/mL. Pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 344 | 123
ug/mL
  Anti-1 | 3.41 [3.14 to 3.71] | 0.04 [0.04 to 0.05]
  Anti-4 | 4.00 [3.67 to 4.35] | 5.35 [4.66 to 6.15]
  Anti-5 | 4.52 [4.24 to 4.83] | 0.07 [0.06 to 0.08]
  Anti-6B | 1.40 [1.24 to 1.58] | 2.07 [1.75 to 2.44]
  Anti-7F | 4.08 [3.77 to 4.41] | 0.03 [0.03 to 0.04]
  Anti-9V | 3.39 [3.09 to 3.71] | 5.09 [4.34 to 5.96]
  Anti-14 | 5.54 [5.02 to 6.12] | 8.51 [7.27 to 9.95]
  Anti-18C | 5.80 [5.17 to 6.52] | 5.13 [4.31 to 6.11]
  Anti-19F | 7.41 [6.67 to 8.23] | 2.77 [2.45 to 3.13]
  Anti-23F | 1.96 [1.75 to 2.19] | 3.94 [3.26 to 4.77]

6. Secondary Outcome: Anti-PD Antibody Concentration
Description: Concentration of anti-PD antibody given as GMC expressed in EL.U/mL.
Time Frame: One month after administration of 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 344 | 123
EL.U/mL | 1622.4 [1500.8 to 1754.0] | 88.2 [74.7 to 104.0]

7. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes
Description: Concentration of cross-reactive pneumococcal serotypes 6A and 19A in ug/mL.
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 344 | 123
ug/mL
  Anti-6A | 0.38 [0.33 to 0.44] | 0.48 [0.36 to 0.63]
  Anti-19A | 0.29 [0.25 to 0.33] | 0.12 [0.10 to 0.14]

8. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Pneumococcal Cross-reactive Serotypes
Description: The results were presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. In this assay the cut-off value for opsonophagocytic activity against pneumococcal cross-reactive serotypes 6A and 19A was defined as >= 8.
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 162 | 60
subjects
  Opsono-6A (N=158; 60) | 134 | 54
  Opsono-19A (N= 162; 60) | 53 | 7

9. Secondary Outcome: Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentrations
Description: Concentration of anti-PRP antibody given as GMC in ug/mL.
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 175 | 60
ug/mL | 20.131 [16.775 to 24.158] | 11.844 [8.542 to 16.424]

10. Secondary Outcome: Number of Subjects With Seroprotection Status Against PRP
Description: Seroprotection status is defined as anti-PRP antibody concentrations above 0.15 ug/mL and above 1.0 ug/mL
Time Frame: One month after the administration of the 3rd vaccine dose of the pneumococcal conjugate vaccine
Population: as for outcome 3
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 175 | 60
subjects
  Above 0.15 | 175 | 60
  Above 1.0 | 173 | 58

11. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: Within 4 days after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 371 | 129
subjects
  Pain | 210 | 72
  Redness | 252 | 84
  Swelling | 182 | 69

12. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever, irritability and loss of appetite.
  Fever was defined as axillary temperature >= 37.5 degrees Celsius.
Time Frame: Within 4 days after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 371 | 129
subjects
  Drowsiness | 212 | 65
  Fever | 113 | 33
  Irritability | 293 | 99
  Loss of Appetite | 177 | 66

13. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Time Frame: Within 31 days after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 374 | 129
subjects | 213 | 62

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Following the administration of the first dose of the study vaccines throughout the entire study period up to study month 5
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Number; unit: subjects
Arm/Group | Synflorix Group | Prevenar Group
Number analyzed (Participants) | 374 | 129
subjects | 56 | 9

ADVERSE EVENTS:
Time Frame: Up to study Month 5
Description: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Arm/Group | Synflorix Group | Prevenar Group
Serious Adverse Events (participants affected / at risk) | 56/374 | 9/129
Other Adverse Events (participants affected / at risk) | 357/374 | 124/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Group (N=374) | Prevenar Group (N=129)
Bronchiolitis (Infections and infestations) | 22 | 1
Gastroenteritis (Infections and infestations) | 8 | 3
Urinary tract infection (Infections and infestations) | 9 | 1
Pneumonia (Infections and infestations) | 4 | 1
Croup infections (Infections and infestations) | 2 | 1
Intussusception (Gastrointestinal disorders) | 2 | 1
Meningitis aseptic (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 3 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0
enteritis (Gastrointestinal disorders) | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Otitis media acute (Infections and infestations) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Exanthema subitum (Infections and infestations) | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Herpangina (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1
Meningitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
rhinitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Group (N=374) | Prevenar Group (N=129)
Pain (General disorders) | 210 | 72
Redness (General disorders) | 252 | 84
Swelling (General disorders) | 182 | 69
Drowsiness (General disorders) | 212 | 65
Fever (General disorders) | 113 | 33
Irritability (General disorders) | 293 | 99
Loss of appetite (General disorders) | 177 | 66
Upper respiratory tract infection (Infections and infestations) | 44 | 16
Nasopharyngitis (Infections and infestations) | 42 | 16
bronchiolitis (Infections and infestations) | 20 | 4
Pharyngitis (Infections and infestations) | 23 | 6
Bronchitis (Infections and infestations) | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.